CLINICAL TRIAL: NCT04712773
Title: Comparison of the Nociception Monitoring Devices During Cardiac Surgery.
Acronym: SYDNOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kuopio University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Kuopio University Hospital
Record Dates: First submitted 2020-12-21; First posted 2021-01-15 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Surgery
Keywords: cardiac surgery; pain; nociception
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cardiac surgery patients (Other): Patients scheduled for elective cardiac surgery (CABG or valve surgery).
  Interventions: Device: PMD-200 monitor; Device: Surgical Pleth Index monitor

INTERVENTIONS:
Device: PMD-200 monitor — Patient is connected to non-invasive PMD-200 monitor, measuring Nociception Level
Device: Surgical Pleth Index monitor — Patient is connected to non-invasive monitor measuring Surgical Pleth Index

SUMMARY:
The purpose of this study is to compare the values of Surgical Pleth Index (SPI) and Nociception Level Index (NOL) measured simultaneously during cardiac surgery.

DETAILED DESCRIPTION:
Participants are given oral and written information about the course of the trial, associated risks and benefits and about the handling of the personal data on the day before the surgery by one of the investigators. Participants are also given written information about patient's rights and insurance, the aim of the trial and its course. 40 adult cardiac surgery patients will be recruited for the study. NOL and SPI values will be measured during the cardiac surgery procedure. All patients receive oral premedication and standardized anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* coronary artery disease of heart valve disorder qualified for the surgical treatment
* participant understands the course of the trial and its aim
* participant has given informed written consent

Exclusion Criteria:

* participant has not given consent
* neurological or psychical disorders (psychiatric medication)
* dementia
* alcohol or substance abuse
* central nervous system medication (medication for epilepsy or neuropathic pain)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-03-01 (Actual)

PRIMARY OUTCOMES:
SPI values measured at several timepoints during cardiac surgery | Values are measured during the course of the cardiac surgery procedure
  SPI (Surgical Pleth Index) - index measuring nociceptive response based on pulse and pulse amplitude.
NOL values measured at several timepoints during cardiac surgery | Values are measured during the course of the cardiac surgery procedure
  NOL (Nociception Level Index) - nociception index based on heart rate and its changes, pulse wave amplitude, skin impedance and its changes, temperature and their variations

CONTACTS AND LOCATIONS:
Overall Officials: Tadeusz Musialowicz, PhD, MD, Study Director — Kuopio University Hospital, Department of Anesthesiology and Intensive Care
Locations (1):
- Kuopio University Hospital, Kuopio, Northern Savonia, Finland

IPD SHARING:
Plan to Share IPD: No